CLINICAL TRIAL: NCT01608282
Title: Capitalizing on the Teachable Moment: the OPEN (Osteoarthritis Physical Activity & Exercise Net) for Improving Physical Activity in Early Knee Osteoarthritis
Brief Title: Internet Intervention to Improve Physical Activity in Early Knee Osteoarthritis
Acronym: OPEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to reach recruitment target
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Simon Fraser University (Other); Arthritis Research Centre of Canada (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H12-00493
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Arthritis; Knee; Exercise; Physical Activity; Web-based
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPEN Intervention Group (Experimental): Intervention group participants will receive an email prompt to access the OPEN website every two weeks for the first three months, with a short message about the ongoing projects at the Arthritis Research Centre of Canada. The OPEN website will remain accessible throughout the study, but no further prompting emails will be sent after Month 3. In addition, they will receive an education pamphlet produced by The Arthritis Society containing information about osteoarthritis, physical activity and other treatments.
  Interventions: Behavioral: OPEN website
- Control Group (No Intervention): Control group participants will receive, by email, the same Arthritis Society pamphlet as the Intervention group. Participants will also receive, by email, the same short message about the ongoing projects at the Arthritis Research Centre of Canada, every two weeks for the first three months (i.e. the same schedule as the intervention group receiving the prompting email so that the number of contacts is equal in both groups), but without the prompting to use the OPEN website.

INTERVENTIONS:
Behavioral: OPEN website — The OPEN website includes interactive modules that allow users to prioritise their daily activities, set goals and find venues where they can participate in different types of activities according to their preferences and the local availability
  Arms: OPEN Intervention Group

SUMMARY:
OPEN (Osteoarthritis Physical Activity and Exercise Net) is a website created based on a well developed behavioural theory. This intervention is developed for people with early knee osteoarthritis (OA) who have been sedentary. The investigators aim to engage these individuals to become physically active at a time when their joint symptoms tend to be mild. The primary goal of this proof-of-concept randomized controlled trial is to determine if the OPEN website plus an information pamphlet about OA will improve participation in physical activity in persons with early knee OA, compared to those who receive only the pamphlet.

DETAILED DESCRIPTION:
Being physically active has been shown to reduce pain, improve quality of life and potentially reduce joint damage. However, our recent survey in British Columbia found only 1 in 4 people with mild osteoarthritis symptoms (pain; stiffness) met the recommended level of physical activity. Research in people without arthritis shows that web-based tools can increase walking behaviour, but none of these tools are designed with the needs of people with arthritis in mind. Research in other chronic diseases has found that people are more likely to quit smoking shortly after the diagnosis of a smoking-related disease. Thus, the diagnosis of osteoarthritis presents an ideal 'teachable moment' to engage those who have been sedentary to become physically active.

This project will address the Research Question: Can an interactive website increase physical activity in people with previously undiagnosed knee OA and those with a diagnosis of knee OA with no contraindication for being physically active? We have created a website, called OPEN (Osteoarthritis Physical Activity & Exercise Net), based on a well developed behavioural theory. A total of 252 sedentary people with knee osteoarthritis will be recruited in British Columbia to test the website. Half of them will be assigned to use the OPEN website for 3 months and will receive an education pamphlet produced by The Arthritis Society; the other half will only receive the pamphlet. During the test period, participants will complete an online questionnaire at 0, 3 and 6 months to allow us to follow changes in physical activity, knee symptoms and outcomes related to their motivation to become physically active. In addition,Participants will be stratified by OA diagnosis (having previously undiagnosed OA, as identified by a validated questionnaire, versus having a knee OA diagnosis). participants from Metro Vancouver who have previously undiagnosed knee OA will complete an aerobic fitness test administered by a blind assessor. Changes between the two groups will be compared.

Our project directly targets physical inactivity at a time when the joint damage tends to be mild, and when people are more motivated to adopt a healthy behaviour. If the OPEN is found to be effective in improving physical activity, it opens further opportunities to promote early diagnosis and to implement lifestyle interventions.

ELIGIBILITY:
Inclusion Criteria:

* Have felt pain/discomfort in or around the knee during the previous year that lasted more than 28 separate or consecutive days.
* Are 50 years or older.
* Have not been physically active regularly (meaning, you have not participated in moderate intensity activities more than 90 minutes a week) in the past six months.
* Have access to the internet.
* Live in British Columbia.

Exclusion Criteria:

* Have physician diagnosis of rheumatoid arthritis, psoriatic arthritis, gout, ankylosing spondylitis, polymyalgia rheumatica, connective tissue diseases or fibromyalgia.
* Have a history of using disease-modifying anti-rheumatic drugs (DMARD) or gout medications.
* Have had total knee replacement surgery or currently being considered for.
* Have had any knee surgery within the past four months.
* Have had acute injury to the knee in the past six months.
* Have been using medication that may impair physical activity tolerance (e.g., beta blockers)
* Are at other risks from exercising as identified by the Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Modified Minnesota Leisure Time Physical Activity Questionnaire (MLTPAQ). | Change from baseline in levels of physical activity at 3 months and 6 months
  Proportion of participants meeting the American College of Sports Medicine physical activity recommendation of 150 minutes or more of weekly physical activity (moderate or heavy intensity).

SECONDARY OUTCOMES:
Knee Injury and OA Outcome Score (KOOS). | Change from baseline in knee pain, stiffness, daily activity, sports/recreation and quality of life at 3 months and 6 months
  The KOOS consists of five subscales: knee pain, stiffness, daily activity, sports/recreation, and quality of life.
Rhode's 7-point Likert-type Theory of Planned Behaviour questionnaire | Change from baseline in motivation for physical activity at 3 months and 6 months
  Motivation for physical activity will be measured with Rhode's 7-point Likert-type Theory of Planned Behaviour (TPB) questionnaire. It consists of 16 items measuring all components of the TPB model, including behavioural, normative and control beliefs.
Aerobic fitness (V02Peak) | Change from baseline in aerobic fitness at 3 months and 6 months
  A sub-sample of participants (n=40) will undergo a submaximal aerobic fitness test at baseline, 3 months and 6 months. Aerobic fitness will be predicted by extrapolating the heart rate and oxygen update responses to three submaximal exercise stages.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — University of British Columbia and Arthritis Research Centre
Locations (1):
- Arthritis Research Centre, Richmond, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li LC, Lineker S, Cibere J, Crooks VA, Jones CA, Kopec JA, Lear SA, Pencharz J, Rhodes RE, Esdaile JM. Capitalizing on the teachable moment: osteoarthritis physical activity and exercise net for improving physical activity in early knee osteoarthritis. JMIR Res Protoc. 2013 May 9;2(1):e17. doi: 10.2196/resprot.2553. PMID 23659903
- See also: OPEN project - Arthritis Research Centre of Canada — http://www.arthritisresearch.ca/top-menu-research-current/research-current/274-osteoarthritis-physical-activity-a-exercise-net.html?catid=64%3Aoa-current-research